CLINICAL TRIAL: NCT02925429
Title: The PostNAPS Study: Food Insecurity As A Major Determinant of Poor Nutritional and Psychosocial Health Outcomes Among HIV-Infected and -Uninfected Lactating Women and Their Infants in Gulu, Northern Uganda.
Brief Title: PostNAPS: FI, Nutrition, and Psychosocial Health Among Women of Mixed HIV Status and Their Infants in Gulu, Uganda
Acronym: PostNAPS
Status: Completed | Type: Observational
Sponsor: Northwestern University (Other)
Collaborators: Cornell University (Other); Tufts University (Other); Weill Medical College of Cornell University (Other); Makerere University (Other)
Responsible Party: Principal Investigator, Sera Young, Associate Professor, Northwestern University
Other Study IDs: 1302003634
Record Dates: First submitted 2016-10-03; First posted 2016-10-05 (Estimated); Last update posted 2020-11-13 (Actual); Status verified 2020-11

CONDITIONS: Food Insecurity; HIV; Maternal and Child Health; Nutrition; Psychosocial Health

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
PostNAPs was a continuation of the PreNAPs study. 246 women were enrolled in the postnatal period with the primary scientific objective of determining whether food insecurity was an independent risk factor for poor maternal nutritional or psychosocial outcomes or for sub-optimal infant feeding practices.

ELIGIBILITY:
Inclusion Criteria:

* Postpartum women >18 years of age
* Attended antenatal care at Gulu Regional Referral Hospital
* Participated in the PreNAPS study
* Infants that were born to women participating in the PreNAPS study

Exclusion Criteria:

* Women <18 years of age
* Women not participating in the PreNAPS study

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Postpartum women >18 years of age of mixed HIV status who had attended antenatal care at Gulu Regional Referral Hospital in Gulu, Uganda and had participated in the PreNAPS longitudinal observational cohort study and their infants.
Sampling Method: Non-Probability Sample
Enrollment: 246 (Actual)
Dates: Start 2013-05; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Impacts of food insecurity (IFIAS) on maternal and infant health indicators (i.e. changes in body composition, hemoglobin, morbidity, etc.) among lactating women of mixed-HIV status and their infants in Gulu, Uganda | Approximately 1 year
  Explore the underlying mechanisms and impacts of food insecurity (using the Individual Food Insecurity Access Scale (IFIAS)) on body composition changes (weight in kg, bioelectrical impedance analysis (among women), skin folds, MUAC), morbidity (malaria, diagnoses or symptoms of fever, typhoid, diarrhea, etc.), micronutrient status (hemoglobin), and other health indicators among women of mixed-HIV status and their infants in Gulu, Uganda.

SECONDARY OUTCOMES:
Impacts of food insecurity (IFIAS) and maternal depression (CES-D) on maternal folate levels among women of mixed-HIV status in Gulu, Uganda. | Approximately 1 year
  Describe the relationship between food insecurity (IFIAS) and maternal depression (CES-D) on maternal folate levels and assess if these relationships are modified by maternal HIV status.
Impacts of food insecurity (IFIAS) and maternal depression (CES-D) on maternal B12 levels among women of mixed-HIV status in Gulu, Uganda. | Approximately 1 year
  Describe the relationship between food insecurity (IFIAS) and maternal depression (CES-D) on maternal B12 levels and assess if this relationship is modified by HIV status.
Impacts of food insecurity (IFIAS) and maternal depression (CESD) on infant feeding among women of mixed-HIV status in Gulu, Uganda | Approximately 1 year
  Explore the impacts of food insecurity (IFIAS) and maternal depression (CESD) on infant feeding (breastfeeding, introduction of complimentary foods, infant dietary diversity).
Changes in food insecurity (IFIAS) within the first year of delivery among women of mixed-HIV status in Gulu, Uganda | Approximately 1 year
  Measure changes in the prevalence and severity of food insecurity from delivery to approximately 1 year postpartum among women of mixed-HIV status in Gulu, Uganda.

CONTACTS AND LOCATIONS:
Overall Officials: Sera L Young, MA, PhD, Principal Investigator — Northwestern University; Barnabas K Natamba, MPH, PhD, Principal Investigator — Michigan State University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lane CE, Widen EM, Collins SM, Young SL. HIV-Exposed, Uninfected Infants in Uganda Experience Poorer Growth and Body Composition Trajectories than HIV-Unexposed Infants. J Acquir Immune Defic Syndr. 2020 Oct 1;85(2):138-147. doi: 10.1097/QAI.0000000000002428. PMID 32604132
- [Derived] Boateng GO, Martin SL, Tuthill EL, Collins SM, Dennis CL, Natamba BK, Young SL. Adaptation and psychometric evaluation of the breastfeeding self-efficacy scale to assess exclusive breastfeeding. BMC Pregnancy Childbirth. 2019 Feb 18;19(1):73. doi: 10.1186/s12884-019-2217-7. PMID 30777020
- [Derived] Boateng GO, Martin SL, Collins SM, Natamba BK, Young SL. Measuring exclusive breastfeeding social support: Scale development and validation in Uganda. Matern Child Nutr. 2018 Jul;14(3):e12579. doi: 10.1111/mcn.12579. Epub 2018 Jan 22. PMID 29356347
- [Derived] Widen EM, Collins SM, Khan H, Biribawa C, Acidri D, Achoko W, Achola H, Ghosh S, Griffiths JK, Young SL. Food insecurity, but not HIV-infection status, is associated with adverse changes in body composition during lactation in Ugandan women of mixed HIV status. Am J Clin Nutr. 2017 Feb;105(2):361-368. doi: 10.3945/ajcn.116.142513. Epub 2017 Jan 4. PMID 28052888